CLINICAL TRIAL: NCT02075788
Title: Millet Products Study - Investigation of Glycemic Index and Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Bunge Global Innovation Incorporated (Unknown)
Responsible Party: Principal Investigator, Amanda Wright, Ph.D., Associate Professor, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 13AP004
Record Dates: First submitted 2014-02-26; First posted 2014-03-03 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Hyperglycemia; Lack of Satiety
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Commercial white bread (Placebo Comparator): All product servings will provide 50 g of available carbohydrate and will be consumed by participants within 10 minutes.
  Interventions: Other: Commercial white bread
- Millet based products (porridge etc.) (Experimental): All product servings will provide 50 g of available carbohydrate and will be consumed by participants within 10 minutes.
  Interventions: Other: Millet based products (porridge etc.)
- Corn based products (porridge etc.) (Active Comparator): All product servings will provide 50 g of available carbohydrate and will be consumed by participants within 10 minutes.
  Interventions: Other: Corn based products (porridge etc.)

INTERVENTIONS:
Other: Commercial white bread
  Arms: Commercial white bread
Other: Corn based products (porridge etc.)
  Arms: Corn based products (porridge etc.)
Other: Millet based products (porridge etc.)
  Arms: Millet based products (porridge etc.)

SUMMARY:
The purpose of this study is to investigate how millet incorporation into different baked product types influences glycemic response and satiety.

DETAILED DESCRIPTION:
The purpose of this study is to investigate how millet incorporation into different baked product types (i.e. an extruded snack versus a biscuit) influences glycemic response and satiety.

This project will examine the effect of millet, on glycemic response and satiety. To determine the effect of product matrix and processing methods, testing will be done using an extruded snack, porridge, a couscous-like product and a biscuit.

All product servings will provide 50 g of available carbohydrate and will be consumed by participants within 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Men, age 19-40, non-smoking
* Normal fasting plasma glucose (<5.6 mmol/L but not below 3.6 mmol/L)
* Normal glucose tolerance (evaluated by a 75 g oral glucose test, i.e. <7.8 mmol/L but not below 3.6 mmol/L)
* BMI ranging from 18.5 to 29.9 kg/m2

Exclusion Criteria:

* Insulin resistance (IR) will be calculated from fasting glucose and insulin values using the Homeostasis Assessment Model 2 (HOMA2). A HOMA2-IR value of greater than 1.0 will be considered indicative of insulin resistance (Levy J.C. et al. 1998).
* Regular consumption of millet as defined by questionnaire at screening defined as more than 1x per week
* Smoking or use of recreational drugs
* Heavy alcohol use (defined as typically >14 drinks per week or >4 drinks on one occasion)
* Very low fibre consumption as assessed by 24 hour food diary and self-reported fruit/vegetable/whole grain servings.
* Restrained eater as defined by the questionnaire at screening (Three Factor Eating Questionnaire, Stunkard et al.,1985)
* Food neophobic defined by Food Neophobia Scale questionnaire
* Unusual sleep patterns or irregular breakfast consumption
* Recent (i.e. >4 kg in previous 3 months) or intended weight loss or gain
* Food allergies or any life-threatening allergy (food or otherwise)
* Inflammatory bowel disease or other gastrointestinal disorders
* Use of drugs which influence carbohydrate metabolism
* Training or elite athletes
* Inability to adhere to Study Protocols

Ages: 19 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Determination of glycemic index based on collection of capillary plasma glucose | Outcome measures will be assessed at fasting, and postprandially at 15, 30, 45, 60, 90 and 120 minutes

SECONDARY OUTCOMES:
Self reported ratings of satiety | Outcome measures will be assessed at fasting, and postprandially every 30 minutes over 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutraceutical Research Unit, University of Guelph, Guelph, Ontario, Canada